CLINICAL TRIAL: NCT04281550
Title: Supporting Optimal Hydration With Those Living With Dementia in Care Homes
Brief Title: Hydration Care in Dementia Care Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Glenda Cook, Professor of nursing, Northumbria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Think Drink
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This study was a three-phase multi-method design consisting of analysis of the empirical grounds for the hydration intervention, development of a multi-component hydration intervention and a feasibility cluster trial of the intervention. The first phase constituted of a survey of care homes, a systematic review-informed review of previous literature and collection of professional perspectives. Second phase was the development the intervention through five workshop events. Finally, the feasibility phase compared 6 intervention homes and 5 control homes in North East England, over a 3-month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Think drink intervention (Experimental): The Think Drink multicomponent hydration intervention was introduced into the intervention group care homes through a staff workshop.
  Interventions: Other: Think Drink

INTERVENTIONS:
Other: Think Drink — The Think Drink Guide that had three interacting components. The 'policy' component was directed at the governance of the care home, whereas 'practice' components were directed at hydration procedures and processes, and 'educational' components that provided learning resources for care home staff to develop knowledge and understanding of hydration care. Think Drink was implemented through a short awareness-raising educational programme and accompanying information booklet detailing a range of practices (including organisational, system and individual practice) designed to encourage hydration.

SUMMARY:
The study aimed to provide evidence of the feasibility of implementing a multi-component intervention for optimising hydration in people with dementia living in care homes.

To undertake a multi method feasibility study to investigate the suitability of methods and outcome measures for future research.

Objectives:

1. Explore personal barriers experienced by people with dementia regarding drinking in care home contexts
2. Explore professional and organisational perspectives of approaches to optimal hydration of residents with dementia and the barriers in everyday practice
3. Develop a multi-component intervention to enhance hydration for residents in collaboration with care home staff, mental health and geriatric specialists, and residents' family
4. Assess the feasibility of implementing the intervention in care homes, and impact on recommended daily intake of fluids
5. Explore the impact of the intervention on daily fluid intake, and designing suitable secondary outcome measures - admission to hospital due to dehydration, falls, laxative use, urinary tract infection, upper respiratory tract infection and skin breakdown.

DETAILED DESCRIPTION:
Previous literature has shown that maintaining adequate hydration levels for residents with dementia can be challenging. This is due to difficulties with swallowing, remembering to get drinks or refusal to drink. Dehydration in people with dementia is a major problem and significant cause of admission to hospital (Bourdel-Marchasson, 2004; Hodgkinson, Evans and Woods, 2003). Despite this, there is limited research into hydration interventions for this population, despite preliminary evidence suggesting the potential benefits of using multi-component interventions (Bunn et al. 2015).

The primary aim of this feasibility study was to establish the feasibility and acceptability of conducting a definitive RCT to evaluate the effectiveness of a multi-component hydration intervention for people living with dementia in nursing care homes compared to usual care.

Secondary aims were to establish:

* Whether the Think Drink intervention can be delivered as planned within nursing care homes for people living with dementia
* If the intervention is acceptable to care home staff
* If it is feasible to recruit and randomise care home sites and participants
* Barriers to the delivery of the Think Drink guide intervention.
* If the outcome measures are feasible to use within a care home setting
* If reliable data can be collected
* A sample size calculation for an RCT. This study was a three-phase multi-method design consisting of analysis of the empirical grounds for the hydration intervention, development of a multi-component hydration intervention and a feasibility cluster trial of the intervention. The first phase constituted of a survey of care homes, a systematic review-informed review of previous literature and collection of professional perspectives. Second phase was the development the intervention through five workshop events. Finally, the feasibility phase compared 6 intervention homes and 5 control homes in North East England, over a 3-month period.

The literature review revealed three articles of limited quality and indicates that there has been limited multi-component interventions promoting hydration care following Bunn et al. (2015)'s original systematic review. Evidence available suggests the importance of combining functional and awareness-raising approaches within multi-component interventions. Professional perspectives also reinforced these findings. This was reflected in the development of the Think Drink Guide that had three interacting components. The 'policy' component was directed at the governance of the care home, whereas 'practice' components were directed at hydration procedures and processes, and 'educational' components that provided learning resources for care home staff to develop knowledge and understanding of hydration care. Think Drink was implemented through a short awareness-raising educational programme and accompanying information booklet detailing a range of practices (including organisational, system and individual practice) designed to encourage hydration.

Key Findings A total of 87 residents were included in the study, 37 as part of the control group and 50 in the intervention group. Overall, 45 care home staff from varied roles participated in interviews to determine the acceptance, barriers and facilitators of the Think Drink Intervention. No significant changes were found in terms of the primary outcome for residents (overall hydration consumption over a seven-day period) following the intervention. However, significant methodological concerns were noted over the use of care home-recorded data, particularly as accurate recording was a key focus of the education component and therefore not influenced in the control homes. It was noted from baseline that resident fluid intakes are inconsistently recorded in terms of detail (e.g. 200mls for a cup of tea offered, with no accurate recording of what was actually drunk). The change to more accurate recording in the intervention homes may have influenced the findings.

Qualitative data found that the training was well-received and valued by staff and care homes, particular in its influence of encouraging more frequent availability of drinks and greater variety of drinks offered. However, organisation and policy changes (such as the development of a specific hydration care plan) were not found. A further methodological concern was the lack of use of the Think Drink booklet, with staff suggesting they would prefer more accessible prompts, such as posters.

An a priori power calculation was carried out for a future trial in this area and, including attrition, it is estimated that 240 total participants would be required in a trial.

Key practice and policy recommendations

* Hydration care requires development for residents with dementia across the care home sector. Although some aspects of this are being achieved within care homes and their respective companies, the findings from this study indicated that several improvements were achieved following implementation of the Think Drink intervention. It is recommended that practice and service developments to hydration care continue to be promoted.
* Analysis of existing care planning processes indicates that hydration is not given a high enough priority, and where attention is given it often focuses on functional aspects of hydration care. More detailed information on cognitive issues or personal strategies for supporting hydration in individual residents could provide benefits in the future, particularly considering high levels of staff turnover in this area and a potential need for healthcare partners to access quick and accurate information about residents.
* An important feature of the Think Drink guide was capturing hydration practices that are implemented in care homes in 5 domains - assessment of hydration norms and problems; hydration support and encouragement; drinking activities; drinking conducive environment; drinking equipment. The researchers recommend that further consideration is given to building on this range of hydration practices, and these aspects of hydration care should be incorporated into care home policy and care home commissioning processes.
* Prior to future research further development of the format and presentation of the Think Drink practices domains, and related resources, such as posters, hydration apps or screensavers that can be displayed throughout a care home, to enable care home staff to raise their awareness of different approaches to hydration care and adopt these in their practice is required.
* The implementation of Think Drink in care homes requires a flexible approach that is tailored to the care home setting. Care home-wide approaches (such as ordering a wide variety of drinks and beverages), ensuring all staff across all care home departments are competent to provide hydration care education (through inclusion of hydration education in induction programmes), and cascade models to promote excellence in hydration practice within a care home, should all be considered.
* Hydration education was an important part of implementing Think Drink in care homes. The researchers recommend that care home staff receive hydration education, both during induction to working in a care home and through ongoing regular updates to contribute to proficiency in hydration care of residents.
* Hydration education should also be available to commissioners so that they can contract and carry out quality inspection visits with understanding of the hydration requirements of residents and the challenges that care home staff experience in supporting residents to drink sufficient fluid.
* The importance of accurate fluid recording should be included in hydration education for care home staff. Improvement in this aspect of practice will support care planning, implementation of effective interventions for those identified as having inadequate fluid intake, and communication with healthcare professionals when residents are referred to primary care and out of hours services due to deteriorating health.

Research recommendations

* This was a feasibility study with the purpose of exploring issues of recruitment, testing the intervention and appraising outcome measurement tools. A recommendation for future research would be to increase the implementation period of Think Drink to 6 months to see if the short-term changes in hydration practice is maintained over time. This may require a larger scale study, however, due to high levels of participant attrition that is expected.
* The findings highlight that there is poor documentation of hydration care planning and resident fluid intake. Some participating care homes developed novel approaches to improve the accuracy of fluid intake. The researchers would recommend further research to assess the feasibility of implementing these practices in other care home settings.
* There was difficulty in recruiting care homes to the feasibility study that involved implementation of Think Drink and data collection over a 3-month period. In future research the timeframe for recruiting homes should account for lengthy recruitment processes.
* The results demonstrate that there is a high level of attrition of care home residents and this should be considered when planning future research and in calculation of sample sizes.
* Robustness of the data collected and outcome measures is a key consideration in the testing of any intervention. This feasibility study highlighted inaccuracies in the measurement of fluid intake and in any future study it is recommended that this is taken into consideration in future research and that this is undertaken by research staff. If research staff are present in care homes that provide services for people with dementia this could be disruptive and distressing for residents, hence the research methodology adopted in future research should enable researchers to participate in care whilst undertaking data collection. This will impact significantly on the funding required to undertake this type of research.

ELIGIBILITY:
Inclusion Criteria

* must be a care home resident
* assent for participation is provided by their surrogate decision maker
* must be able to drink oral fluids

Exclusion Criteria

* unable to drink oral fluids
* receiving end of life care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Fluid intake | 6 months
  Change in proportion of the resident population with higher daily fluid intake
Fluid intake 2 | 6 months
  Change in mean fluid intake of drinks that are a) offered and b) consumed

SECONDARY OUTCOMES:
Hydration care plan | 6 months
  Change in residents hydration care plan
Hospital admission | 6 months
  Admission to hospital with diagnosis of dehydration
Death | 6 months
  Death following diagnosis of dehydration
Referral to GP | 6 months
  Change in number of calls to OOH GP services for low fluid intake
UTI | 6 months
  Change in number of residents with UTI
Falls | 6 months
  Change in number of falls
Respiratory tract infection | 6 months
  Change in number of upper respiratory tract infections
Sample attrition | 6 months
  Sample attrition

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Cook, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No